CLINICAL TRIAL: NCT06012695
Title: A Phase Ib/II, Open-label Study of NBM-BMX As Monotherapy or in Combination with Radiotherapy and Temozolomide in Subjects with Solid Tumors or Newly Diagnosed Glioblastoma
Brief Title: NBM-BMX Administered Orally to Patients with Solid Tumors or Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novelwise Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBM-BMX-003
Record Dates: First submitted 2023-08-11; First posted 2023-08-25 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasm; Malignant Neoplasm of Brain
MeSH Terms: conditions — Neoplasms; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- monotherapy in advanced solid tumors (Experimental): Subjects with advanced solid tumors will be treated with NBM-BMX monotherapy at different dose levels depending on the order of their enrollment.
  Interventions: Drug: NBM-BMX Capsule
- combination therapy in newly diagnosed glioblastoma (Experimental): Subjects with newly diagnosed glioblastoma will be treated with NBM-BMX at different dose levels in combination with the standard of care treatment (concomitant RT/TMZ followed by adjuvant TMZ). In the expansion study, Subjects will be treated with NBM-BMX at the recommended Phase 2 dose (RP2D) in combination with RT/TMZ.
  Interventions: Drug: NBM-BMX Capsule; Drug: Temozolomide; Radiation: Standard radiotherapy

INTERVENTIONS:
Drug: NBM-BMX Capsule — Each capsule contains 100 mg of the active ingredient.
Drug: Temozolomide — TMZ will be administered orally at a 75 mg/m2 dose daily during concomitant therapy. In the maintenance period, days 1-5 of each cycle will be administered 150-200 mg/m2.
  Other Names: Temodal® Capsules
  Arms: combination therapy in newly diagnosed glioblastoma
Radiation: Standard radiotherapy — A total dose of 60 Gy will be administered in 6 weeks.
  Arms: combination therapy in newly diagnosed glioblastoma

SUMMARY:
NBM-BMX is an orally available new chemical entity to inhibit histone deacetylases 8 (HDAC8) activity specifically, being developed as a potential anti-cancer therapeutic by NatureWise. This study aims to evaluate the safety, pharmacokinetics, and preliminary efficacy of NBM-BMX as monotherapy in subjects with advanced solid tumors or combination with the standard of care treatment in subjects with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
This is a multi-center, open-label, 2-arm, phase Ib/II study to evaluate the safety, pharmacokinetics, and preliminary efficacy of NBM-BMX as monotherapy in the treatment of solid tumors (Arm A) or in combination with radiotherapy/temozolomide in the treatment of glioblastoma (Arm B).

Arm A consists of dose escalation cohorts in subjects with advanced solid tumors who will be treated with NBM-BMX monotherapy at different dose levels. Arm B consists of dose escalation cohorts (Phase Ib) and expansion cohorts (Phase II) in subjects with newly diagnosed glioblastoma (GBM). Subjects will be treated with NBM-BMX at different dose levels in combination with the first-line standard of care treatment (i.e., concomitant Radiotherapy (RT)/TMZ followed by adjuvant TMZ) in Phase Ib. After the recommended Phase 2 dose (RP2D) is determined in Phase Ib, additional subjects will be enrolled and treated at the RP2D to evaluate the efficacy of NBM-BMX combination therapy.

ELIGIBILITY:
Inclusion Criteria:

Arm A (advanced solid tumors)

1. Having signed and dated the informed consent form.
2. Females or males > 18 years old.
3. Histologically or cytologically confirmed advanced solid tumors refractory to standard of care therapy, or for which no standard of care therapy is available.
4. Disease that is measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Response Assessment in Neuro-Oncology (RANO) criteria (for CNS tumors).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
6. Adequate organ function as defined by the following criteria:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 3 × upper limits of normal (ULN), unless liver metastases present, then ≤ 5 × ULN
   2. Total serum bilirubin ≤ 1.5 × ULN unless bilirubin elevation is related to Gilbert's Syndrome for which bilirubin ≤ 3 × ULN
   3. Absolute neutrophil count (ANC) ≥ 1,000/μL
   4. Platelets ≥ 75,000/μL
   5. Hemoglobin ≥ 8.0 g/dL
   6. Non-indexed estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m2 × BSA (m2)/1.73.

   Transfusion is not allowed to meet entry criteria.
7. QTcF ≤ 480 msec
8. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Arm B (newly diagnosed GBM)

1. Having signed and dated the informed consent form.
2. Females or males > 18 years old.
3. Newly diagnosed, histologically confirmed glioblastoma, non-resectable, partially resected or resected.
4. Karnofsky performance status (KPS) ≥ 60 at screening and before the initiation (Day 1) of concomitant therapy.
5. Disease that is measurable or evaluable as defined by Response Assessment in Neuro-Oncology (RANO) criteria.
6. Adequate organ function as defined by the following criteria:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 3 × upper limit of normal (ULN), unless liver metastases present, then ≤ 5 × ULN
   2. Total serum bilirubin ≤ 1.5 × ULN unless bilirubin elevation is related to Gilbert's Syndrome for which bilirubin ≤ 3 × ULN
   3. Absolute neutrophil count (ANC) ≥ 1,500/μL
   4. Platelets ≥ 100,000/μL
   5. Hemoglobin ≥ 8.0 g/dL
   6. Non-indexed estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 × BSA (m2)/1.73.

   Transfusion is not allowed to meet entry criteria.
7. QTcF ≤ 480 msec
8. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

Arm A (advanced solid tumors)

1. Systemic anti-cancer treatment (investigational or approved) within 28 days or 5 half-lives of that drug (whichever is shorter) of the first dose of NBM-BMX.
2. Curative radiation therapy within 28 days or palliative RT within 7 days of the first dose of NBM-BMX.
3. Currently taking strong inhibitors (e.g., gemfibrozil) or inducers of CYP2C8.
4. Any of the following within 6 months of the first dose of NBM-BMX: pulmonary embolism events, deep vein thrombosis (DVT) events, myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
5. A positive test for hepatitis B (HBsAg) and/or hepatitis C (anti-HCV antibody), unless the HBV DNA level and/or HCV RNA level is below the limit of detection.
6. Known history of human immunodeficiency virus (HIV) infection.
7. Men and women of childbearing potential who are unwilling to use highly effective contraceptive methods during the study period.

   Highly effective contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, surgical sterilization or a partner who is sterile.
8. Females who are pregnant or breastfeeding.
9. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgement of the investigator and/or sponsor, excess risks associated with study participation or study drug administration.

Arm B (newly diagnosed GBM)

1. Prior systemic therapy (including Gliadel wafer implant), immunotherapy, investigational agents, or radiotherapy for glioblastoma.
2. Currently taking strong inhibitors (e.g., gemfibrozil) or inducers of CYP2C8.
3. Corticosteroid use of > 8 mg/day dexamethasone or equivalent within 5 days before the first dose of NBM-BMX.
4. A history of hypersensitivity reaction to temozolomide or dacarbazine.
5. Any of the following within 6 months of the first dose of NBM-BMX: pulmonary embolism events, deep vein thrombosis (DVT) events, myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
6. A positive test for hepatitis B (HBsAg) and/or hepatitis C (anti-HCV antibody), unless the HBV DNA level and/or HCV RNA level is below the limit of detection.
7. Known history of human immunodeficiency virus (HIV) infection. Note: HIV testing is not required.
8. Men and women of childbearing potential who are unwilling to use highly effective contraceptive methods during the study period and for at least 6 months after the final dose of temozolomide.

   Highly effective contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, surgical sterilization or a partner who is sterile.
9. Female who are pregnant or breastfeeding.
10. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgement of the investigator and/or sponsor, excess risks associated with study participation or study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
[Arm A, Phase Ib] Frequency of dose-limiting toxicity (DLT) at each dose level | up to 28 days
  To determine the maximum tolerated dose (MTD) for NBM-BMX monotherapy in subjects with advanced solid tumors, toxicities will be graded according to the National Cancer Institute Common Terminology.
[Arm B, Phase Ib] Frequency of dose-limiting toxicity (DLT) at each dose level | up to 10 weeks
  To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) for NBM-BMX in combination with RT and TMZ in subjects with newly diagnosed GBM, toxicities will be graded according to the National Cancer Institute Common Terminology.
[Arm B, Phase II] Progression-free survival rate at 6 months (PFS6) | up to 6 months
  To assess the preliminary efficacy of NBM-BMX in combination with RT and TMZ in subjects with newly diagnosed GBM, the investigators will evaluate anti-tumor activity using RANO criteria.

SECONDARY OUTCOMES:
Frequency, types, severity, and relationship to NBM-BMX of adverse events (AEs) | up to 28 days
  The severity of AEs will be graded using NCI CTCAE Version 5.0 by the investigator.
Preliminary assessment of anti-tumor activity by response evaluation criteria | at least 8 weeks
  Tumor response and progression will be assessed using the RECIST v1.1 or Response Assessment in Neuro-Oncology (RANO) criteria.
Area under the plasma concentration versus time curve (AUC) of NBM-BMX | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Blood samples will be collected at each pre-specified time point for measuring concentrations of NBM-BMX in plasma using a validated bioanalytical method.
Peak plasma concentration (Cmax) of NBM-BMX | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Blood samples will be collected at each pre-specified time point for measuring concentrations of NBM-BMX in plasma using a validated bioanalytical method.
Time to maximum plasma concentration (Tmax) of NBM-BMX | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Blood samples will be collected at each pre-specified time point for measuring concentrations of NBM-BMX in plasma using a validated bioanalytical method.
Terminal elimination half-life (T1/2) of NBM-BMX | Day 1, 8 and 15 for Cycle 1 only (each cycle is 28 days)
  Blood samples will be collected at each pre-specified time point for measuring concentrations of NBM-BMX in plasma using a validated bioanalytical method.

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Linkou Chang-Gung Memorial Hospital, Taoyuan